CLINICAL TRIAL: NCT06097559
Title: A Multicenter, Prospective, Non-selection Study for Endometrial Receptivity Analysis Test in Patients With Previous Implantation Failures
Brief Title: International Non-selection Study for ERA® Test in Patients With Previous Implantation Failures
Status: Active, not recruiting | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-ENS-MR-22-05
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Infertility of Uterine Origin; Implantation Failure
Keywords: Infertility; Implantation failure; Uterine microbiome; Preimplantational Genetic Testing for Aneuploidies; Endometrial factor; Window of implantation; Endometrial receptivity; Personalized embryo transfer; Frozen embryo transfer; Endometrial Receptivity Analysis (ERA)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from endometrial fluid and biopsy to analyze the WOI and the endometrial microbiome.
  Provided that the patient (or representative) has granted the corresponding authorization, the endometrial biopsy remnants may be used to continue improving knowledge about diseases that affect infertility in related future studies. These samples will be stored at the Igenomix facilities as part of an Official Biological Sample Collection registered in the name of Dr. Carmen Rubio, Vice President of Genetic Services R&D in Igenomix Research & Development, (reference code of the collection in the National Biobank Registry of the Instituto de Salud Carlos III: C.0007917).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clinical Outcomes in a Receptive Endometrium: Enrolled patients that according to the ERA® report are receptive.
  The only additional intervention that patients will undergo, apart from those already scheduled for their ART, is the collection of an endometrial biopsy and endometrial fluid.
  No drugs will be administered as per the study.
  Interventions: Diagnostic Test: Endometrial fluid and biopsy collection
- Clinical Outcomes in a Non-receptive Endometrium: Enrolled patients that according to the ERA® report have a displaced WOI and are non-receptive.
  The only additional intervention that patients will undergo, apart from those already scheduled for their ART, is the collection of an endometrial biopsy and endometrial fluid.
  No drugs will be administered as per the study.
  Interventions: Diagnostic Test: Endometrial fluid and biopsy collection

INTERVENTIONS:
Diagnostic Test: Endometrial fluid and biopsy collection — The ERA and EMMA test require an endometrial biopsy to be taken at P+5 (after 120±6 hours of exogenous progesterone administration) in a HRT cycle, according to the common clinical practice. On the same day, a sample of endometrial fluid will be aspirated immediately prior to the biopsy.
  Regardless of the endometrial receptivity profile, a subsequent regular FET will be performed within the standard WOI (after 120±6 hours of progesterone exposure) in an HRT cycle following the clinical standard practice.
  Those patients willing to participate in the rescue phase will follow the recommendation of the ERA test for the subsequent pET.
  Groups: Clinical Outcomes in a Receptive Endometrium
Diagnostic Test: Endometrial fluid and biopsy collection — The ERA and EMMA test require an endometrial biopsy to be taken at P+5 (after 120±6 hours of exogenous progesterone administration), according to the common clinical practice. On the same day, a sample of endometrial fluid will be aspirated immediately prior to the biopsy.
  Regardless of the endometrial receptivity profile, a subsequent regular FET will be performed within the standard WOI (after 120±6 hours of progesterone exposure) in an HRT cycle following the clinical standard practice.
  Those patients willing to participate in the rescue phase will follow the recommendation of the ERA test for the subsequent pET. In case of a non-receptive endometrium result, a second EB sample must be collected when indicated by the ERA report. Fluid sample collection will not be repeated in these cases.
  Groups: Clinical Outcomes in a Non-receptive Endometrium

SUMMARY:
Women´s period comprises different hormonal stages, being one of them the stage for maximum receptivity and proper embryo implantation. This stage is named window of implantation (WOI), and is characterized by a specific molecular pattern than can be assessed by the Endometrial Receptivity Analysis (ERA® test), developed by Igenomix. Determining the WOI allows to schedule a personalized embryo transfer (pET) when the endometrium is most receptive for the implantation.

The main objective of the present study is to improve our knowledge on the endometrial factor in an infertile population with previous implantation failures. To do so, a diagnosis of the endometrial receptivity to determine the WOI (ERA®) and the microbiome (EMMA®) of each participant will be performed, assessing its impact on deferred embryo transfers in terms of reproductive outcomes.

Participants will follow their previously programmed IVF/ICSI treatment and, only when one embryo with no major anomalies is reported by PGT-A (Preimplantation Genetic Testing for Aneuploidies), they will be asked to attend to the specific study visit for endometrial fluid and biopsy samples collection. These samples will be used to determine the patient's WOI (ERA®) and endometrial microbiome (EMMA®). The results of neither of the tests will be disclosed to the patient or the doctor, being only used for the study purpose. After this visit, the patient will follow the pre-established schedule for an embryo transfer and pregnancy assessment.

DETAILED DESCRIPTION:
Endometrial receptivity takes place in a self-limited period of time during the endometrial mid-secretory stage. This period, named as window of implantation (WOI), is modulated by molecular changes allowing embryo implantation. The Igenomix group developed a molecular tool able to classify the endometrium based on its transcriptomic profile, the Endometrial Receptivity Analysis (ERA®). This molecular tool analyzes, by next generation sequencing (NGS), the expression of 248 genes related to implantation, coupled to a computational predictor, to identify the specific transcriptomic profile for each endometrial phase. This test has been applied clinically since 2010 to improve clinical implantation, helping to synchronize a viable embryo with a receptive endometrium through the personalized embryo transfer (pET).

Apart from receptivity, there are other approaches to study the impact of the endometrial factor in infertility. One of those is the analysis of the endometrial microbiome (set of microorganisms that live in the endometrium). A reduced presence of certain beneficial microorganisms (mostly, bacteria of the genus Lactobacillus) or even the presence of a pathogenic microbiota in the endometrium could be associated with worse reproductive outcomes, affecting embryo implantation, pregnancy and consequently reducing the number of births. Igenomix has also developed the Endometrial Microbiome Metagenomic Analysis (EMMA®) as a diagnostic method to assess the microbiome content of the endometrium. Both, ERA® and EMMA® analyses, can be performed with a single endometrial tissue sample collected when maximum receptivity is commonly expected.

The main questions this study aims to answer are:

1. If a pET in a specific receptive endometrial transcriptomic profile is related to a higher Ongoing Pregnancy Rate (OPR) (≥ 12 gestational weeks; fetal heartbeat diagnosis) in patients with at least one previous implantation failure. This may help to fine-tune the ERA computational analysis for some specific endometrial receptivity profiles.
2. To identify new potential biomarkers and other factors that, if related with the WOI, could help to predict an optimal embryo implantation.

Once the study is approved by the competent Research Ethics Committee of each center, the recruitment and selection of patients will follow. Every potential participant will be asked to sign the study informed consent. To comply with the study design and the proposed hypothesis, a total number of 738 patients has been estimated, considering a 30% dropout rate.

This is a multicenter, international, competitive, non-selection (prospective cohort) study designed with two phases:

* Non-selection phase (double-blinded design). Participants will follow their previously programmed IVF/ICSI treatment and the resulting embryo/s will be tested for chromosomic anomalies with the Preimplantation Genetic Testing for Aneuploidies (PGT-A) at Igenomix. When at least one euploid/low-range mosaic blastocyst is reported, the patient will be scheduled for the only additional visit related to the study to collect the endometrial fluid and biopsy samples that will be used to determine the patient's WOI (ERA®) and endometrial microbiome (EMMA®). The results of neither of the tests will be disclosed to the patient or the doctor. Therefore, regardless of the endometrial status, the patient will follow the pre-established schedule for a subsequent regular frozen embryo transfer (FET) within the standard WOI (after 120±6 hours of progesterone exposure) in a hormone replacement therapy (HRT) cycle. After the FET, participants will be followed up as routine by their gynecologist.
* Rescue phase (open design). The ERA® test result may be disclosed, under request, to those patients who did not achieve an ongoing pregnancy on the non-selection phase. These results could guide a subsequent personalized euploid/low-range mosaic blastocyst transfer (pET) in a new HRT cycle, when the patient is most receptive.

Data exported from the medical records and source documents will be duly codified to protect the clinical and personal information of patients in accordance with the current legislation on data protection. This information will be exported to an electronic Case Report Form (eCRF). An interim data analysis will be carried out once the 30% of the embryo transfers corresponding to the non-selection phase is achieved. It will help us to assess the enrollment rate, protocol compliance and an early evaluation of the study objectives.

Patient´s participation will comprise an estimated total time of up to 18 months, corresponding to 1 month for the stimulation cycle and PGT-A, 1-2 months for endometrial samples collection, 1-2 months for the embryo transfer and up to 13 months to follow-up the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Study ICF signature.
* Female age between 18 and 41 years (both included).
* IVF/ICSI (own or donated gametes) patients with ≥1 previous failed euploid/low-range mosaic embryo transfer(s) or ≥2 previous failed transfers with non-tested good quality embryos. (ROPA method is allowed).
* ≥1 PGT-A tested euploid/low-range mosaic blastocyst (day 5/6) available to be transferred (SET or DET according to medical recommendation).
* BMI 18.0 - 30.0 Kg/m2.
* Negative serological tests for HIV, HBV, HCV, RPR.

Exclusion Criteria:

* No HRT in the biopsy and/or the embryo transfer cycle.
* Intrauterine device (IUD) carriers within 3 months before sample collection.
* Surrogate pregnancy (in those countries where it is allowed).
* Adenomyosis or any pathological finding affecting the endometrial cavity such as polyps/sub-mucosal myomas, intramural myomas > 4 cm, or hydrosalpinx. (Note: Patients are allowed to participate if the pathology is previously operated at least 3 months before the endometrial samples are obtained).
* Recurrent Pregnancy Loss (RPL ≥2 previous intrauterine miscarriages).
* Active endometritis and salpingitis at the moment of the inclusion.
* Endometriosis stage > I (stages II, III and IV) according to ASRM classification.
* Atrophic endometrium (< 6 mm) in the ERA® and/or embryo transfer cycle.
* Endometrial receptivity test and/or microbiome test done before ICF signature.
* Preimplantation Genetic Testing for Chromosomal Structural Rearrangements (PGT-SR) or Preimplantation Genetic Testing for Monogenic Disorders (PGT-M) concomitant indications.
* DuoStim IVF protocol (double ovarian stimulation and two egg retrievals in the same ovarian cycle).
* Any illness or medical condition that is unstable or which, according to medical criteria, may put at risk the patient's safety and her compliance in the study.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile women scheduled for an in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) cycle with one or more previous failed euploid/low-range mosaic embryo transfer(s) or with two or more previous failed transfers with non-tested good quality embryos, who will receive a transfer of a frozen euploid/low-range mosaic blastocyst (day 5/6) in an HRT cycle.
Sampling Method: Non-Probability Sample
Enrollment: 738 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Refinement of the ERA® computational analysis | At least 12 gestational weeks
  Comparison of the OPR (≥ 12 gestational weeks; fetal heartbeat diagnosis) in patients with receptive endometrium vs displaced WOI in the 1st FET.

SECONDARY OUTCOMES:
Pregnancy rate (PR) in the FET | 2 weeks after the embryo transfer
  Number of patients with positive serum level of β-human chorionic gonadotropin (βhCG > 25 mIU/ml) per embryo transfer. Beta-hCG will be measured at day 12±2 after the embryo transfer.
Implantation rate (IR) in the FET | Up to 4 weeks after the embryo transfer
  Number of gestational sacs observed by vaginal ultrasound divided by the number of embryos transferred.
Biochemical pregnancy rate (BPR) in the FET | 4 weeks after the embryo transfer
  Number of pregnancies diagnosed only by β-hCG detection without a gestational sac visualized by vaginal ultrasound, per number of pregnancies.
Ectopic pregnancy rate (EPR) in the FET | 4-5 weeks after the embryo transfer
  Number of pregnancies outside the uterine cavity, diagnosed clinically, hormonally, by ultrasound, surgical visualization or histopathology, per number of pregnancies.
Clinical miscarriage rate (CMR) in the FET | Up to 22 gestational weeks
  Number of spontaneous pregnancy losses before week 22, in which a gestational sac/s was previously observed, per number of pregnancies.
Ongoing Pregnancy Rate (OPR) in the FET | Over 12 gestational weeks
  Number of pregnancies up to 12 gestational weeks (at least one fetus with a discernible heartbeat diagnosed) achieved per each embryo transfer.
Live Birth Delivery Rate (LBDR) in the FET | 40 gestational weeks
  Number of deliveries that resulted in at least one live birth per embryo transfer. Live birth is defined as the complete expulsion or extraction from a woman of a product of conception after 22 weeks of gestation, which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached.
Pregnancy rate (PR) in the pET | 2 weeks after the embryo transfer
  Number of patients with positive serum level of β-human chorionic gonadotropin (βhCG > 25 mIU/ml) per embryo transfer. Beta-hCG will be measured at day 12±2 after the embryo transfer.
Implantation rate (IR) in the pET | Up to 4 weeks after the embryo transfer
  Number of gestational sacs observed by vaginal ultrasound divided by the number of embryos transferred.
Biochemical pregnancy rate (BPR) in the pET | 4 weeks after the embryo transfer
  Number of pregnancies diagnosed only by β-hCG detection without a gestational sac visualized by vaginal ultrasound, per number of pregnancies.
Ectopic pregnancy rate (EPR) in the pET | 4-5 weeks after the embryo transfer
  Number of pregnancies outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology, per number of pregnancies.
Clinical miscarriage rate (CMR) in the pET | Up to 22 gestational weeks
  Number of spontaneous pregnancy losses before week 22, in which a gestational sac/s was previously observed, per number of pregnancies.
Ongoing Pregnancy Rate (OPR) in the pET | Over 12 gestational weeks
  Number of pregnancies up to 12 gestational weeks (at least one fetus with a discernible heartbeat diagnosed) achieved per each embryo transfer.
Identification of new potential actionable biomarkers for endometrial receptivity | 1-2 months
  Associated genes potentially related with metabolic, inflammatory, and immunological pathways from mRNA ERA® samples.
Clinical reproductive outcomes according to the microbiome profile by the EMMA® test | Up to 40 gestational weeks
  Analysis of the bacterial DNA by next generation sequencing and its possible influence in PR, IR, BPR, EPR, CMR, OPR and LBDR.
Microbiome analysis concordance between endometrial fluid and biopsy | 1-2 months
  Comparison of the EMMA® test results with endometrial biopsy and endometrial fluid
Determination of immune and metabolic changes related to endometrial receptivity | 1-2 months
  Finding of novel underlying mechanisms of impaired endometrium receptivity caused by immune and metabolic alterations
Cost-effectiveness of OP per patient | At least 12 gestational weeks
  Calculation of the cost of pregnancy achievement per patient

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ruiz, MSc, Principal Investigator — Igenomix
Locations (8):
- In Vitro Buenos Aires, Buenos Aires, Buenos Aires, Argentina
- The Fertile Group, Panama City, Panama
- Inmater, San Borja, Lima region, Peru
- Spain (5):
  - Ovoclinic Madrid, Madrid, Madrid
  - Ovoclinic Marbella, Marbella, Málaga
  - URE Centro Gutenberg, Málaga, Málaga
  - Vida Recoletas Sevilla, Seville, Sevilla
  - Vida Recoletas Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No